CLINICAL TRIAL: NCT01437852
Title: An Open-Label, Controlled, Randomized, Multicenter, Dose Escalation Study Evaluating the Safety and Efficacy of StrataGraft® Skin Tissue in Promoting the Healing of the Deep Partial-Thickness Component of Complex Skin Defects as an Alternative to Autografting
Brief Title: StrataGraft® Skin Tissue as an Alternative to Autografting Deep Partial-Thickness Burns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STRATA2011; WFUHS 40269 (Other Grant/Funding Number: AFIRM)
Record Dates: First submitted 2011-09-19; First posted 2011-09-21 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2018-12

CONDITIONS: Skin Wound; Burns; Trauma-related Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- StrataGraft skin tissue (Experimental): All subjects enrolled in this study will receive StrataGraft tissue. Will randomly assign treatment regimens to the two comparable study treatment sites pre-identified as A or B. A sealed randomization envelope will be supplied to the clinical site along with the shipment of clinical tissue. Neither the surgeon nor scrubbed operating room personnel will be informed of the randomization until completion of surgical excision. The treatment sites A or B will be randomized to receive either StrataGraft skin tissue or autograft using a 1:1 ratio.
  Two comparable areas of healthy skin will be pre-identified by the clinical staff as donor sites A or B. The randomization assignment will be identical as that above for the treatment sites. For example, if treatment site A is randomized to receive an autograft, donor site A will be designated the donor site for autografting
  Interventions: Biological: StrataGraft Skin Tissue

INTERVENTIONS:
Biological: StrataGraft Skin Tissue

SUMMARY:
The proposed study is designed as a phase Ib open-label, dose-escalation, multicenter study evaluating the safety, tolerability, and efficacy of StrataGraft skin tissue in promoting the healing of the deep partial-thickness component of complex skin defects. The proposed study population will include patients with 3-49% Total Body Surface Area (TBSA) complex skin defects including a deep partial-thickness component resulting from thermal injury. The study has been designed to focus on the evaluation of safety and tolerability of prolonged exposure to increasing amounts of a single application of StrataGraft skin tissue, while also assessing the potential for StrataGraft tissue to promote healing of the deep partial-thickness component of these complex skin defects as an alternative to donor site harvesting and autografting. Targeted enrollment for this study is up to 30 patients with complex skin defects due to thermal burns which require surgical excision and autografting. Subjects will be sequentially enrolled in two cohorts of increasing treatment area receiving StrataGraft skin tissue that has been stored refrigerated prior to clinical use. A third cohort will receive StrataGraft skin tissue which has been stored cryopreserved and thawed in the operating room just prior to grafting.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-65 years, inclusive
* Written informed consent
* Sufficient healthy skin identified and designated as a donor site in the event that the StrataGraft treatment site requires autografting
* Complex skin defects of 3-49% TBSA requiring excision and autografting
* Total burn may consist of more than one wound area
* Deep partial-thickness thermal burn(s) with total area of 88 to 880 cm2 requiring excision and autografting
* First excision and grafting of treatment sites

Exclusion Criteria:

* Pregnant women and prisoners
* Patients receiving systemic immunosuppressive therapy
* Patients with a known history of malignancy
* Preadmission insulin-dependent diabetic patients
* Patients with concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives
* Expected survival of less than three months
* Participation in the treatment group of an interventional study within preceding 90 days prior to enrollment
* Full-thickness burns will be excluded as treatment sites
* Chronic wounds will be excluded as treatment sites
* The face, head, neck, hands, feet, buttocks, and areas over joints will be excluded as treatment sites
* Treatment sites adjacent to unexcised eschar
* Clinical suspicion of burn wound infection at the anticipated treatment sites

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Stratatech, Inc., a Mallinckrodt Pharmaceuticals Company
Locations (6):
- United States (6):
  - Maricopa Integrated Health Systems, Arizona Burn Center, Phoenix, Arizona
  - University of Colorado Hospital Burn Center, Aurora, Colorado
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - UT-Southwestern Medical Center, Dallas, Texas
  - U.S. Army Institute of Surgical Research, Fort Sam Houston, Texas
  - University of Wisconsin Hospital, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study evaluated the safety and efficacy of StrataGraft skin tissue in promoting the healing of deep partial-thickness burns. Subjects had surgical excision and placement of StrataGraft skin tissue and autograft. The trial was conducted at six clinical sites throughout the United States.
Pre-assignment Details: All subjects were treated with both StrataGraft skin tissue and autograft as part of the intrapatient comparator design. Two comparable excised areas of deep partial-thickness burn per subject were randomized to receive a single application of autograft or StrataGraft skin tissue.
Groups:
- StrataGraft Skin Tissue : Autograft: Two comparable deep partial-thickness burns were excised and randomized to receive StrataGraft skin tissue or autograft.
Period: Overall Study
Arm/Group | StrataGraft Skin Tissue : Autograft
Started | 30
Received StrataGraft Skin Tissue | 30
Received Autograft | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | StrataGraft Skin Tissue : Autograft
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wound Closure of the Treatment Sites at Three Months
Description: Determination of complete wound closure of both treatment sites was evaluated at 3 months.
Time Frame: 3 months
Population: Intent-to-Treat (ITT) Population consisted of all participants who received any amount of StrataGraft skin tissue, regardless of follow-up status. Participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- StrataGraft Skin Tissue: StrataGraft skin tissue is a fully-differentiated tissue which exhibits barrier function comparable to that of intact human skin. StrataGraft consists of an epidermal layer of fully-stratified human keratinocytes growing on a dermal layer which is comprised of human fibroblasts embedded in a collagen matrix. StrataGraft skin tissue is a tough, suturable, meshable tissue product that is manufactured with a surface area of 44 cm2. StrataGraft tissue is not intended to be a patient-specific product but rather to provide an allogeneic skin substitute which reproduces many of the structural and biological properties of normal human skin and is anticipated to serve as a biological wound dressing.
- Autograft: The current standard of care for the management of severe burns and other skin trauma is excision of the necrotic tissue followed by autografting.
Arm/Group | StrataGraft Skin Tissue | Autograft
Number analyzed (Participants) | 29 | 29
Participants | 29 | 29

2. Primary Outcome: Percent Area of the StrataGraft Treatment Site Requiring Autografting by Day 28
Description: The percentage of the treatment site area initially covered with StrataGraft tissue that required autograft by day 28 was determined.
Time Frame: 28 days
Population: ITT Population - consisted of all participants who received any amount of StrataGraft skin tissue, regardless of follow-up status.
Measure: Median (Full Range); unit: Percentage of area
Arm/Group | StrataGraft Skin Tissue
Number analyzed (Participants) | 30
Percentage of area | 0 [0 to 100]

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: All participants who were treated with StrataGraft skin tissue were included in the safety analysis.
Arm/Group | StrataGraft Skin Tissue : Autograft
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StrataGraft Skin Tissue : Autograft (N=30)
Cellulitis (Infections and infestations) | 1 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Impaired healing (General disorders) | 1 (1) — AE considered possibly related to the StrataGraft skin tissue treatment due to inappropriate selection of full-thickness wound that did not meet study inclusion.
Pain (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pneumonia (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Thermal burn (Skin and subcutaneous tissue disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Transplant failure (Skin and subcutaneous tissue disorders) | 2 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Deep vein thrombosis (Vascular disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | StrataGraft Skin Tissue : Autograft (N=30)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Abscess, limb (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Anaemia (Blood and lymphatic system disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Anxiety (Psychiatric disorders) | 3 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — Adverse events (AE) were judged to be possibly related to treatment with StrataGraft skin tissue.
Cardiac failure, congestive (Cardiac disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Cephalohematoma (Injury, poisoning and procedural complications) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Chest pain (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Chills (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Constipation (Gastrointestinal disorders) | 1 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Corneal neovascularization (Eye disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Debridement (Surgical and medical procedures) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Dizziness (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Dyspepsia (Gastrointestinal disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Excoriation (Injury, poisoning and procedural complications) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Eyelid oedema (Eye disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Fluid overload (Metabolism and nutrition disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Fungal infection (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Gastroenteritis (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Gastrointestinal infection (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Gout (Immune system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Graft complication (Injury, poisoning and procedural complications) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Graft infection (Injury, poisoning and procedural complications) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Headache (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Haemorrhoids (Gastrointestinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Herpes simplex (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hyperaesthesia (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypermetabolism (Metabolism and nutrition disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypertension (Vascular disorders) | 3 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypoaesthesia (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypotension (Vascular disorders) | 2 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Ileus (Gastrointestinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Impaired healing (General disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Influenza (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Intestinal functional disorder (Gastrointestinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Joint contracture (Musculoskeletal and connective tissue disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Joint injury (Injury, poisoning and procedural complications) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Keratitis, fungal (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Laceration (Injury, poisoning and procedural complications) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Muscule contracture (Musculoskeletal and connective tissue disorders) | 1 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Nasopharyngitis (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Nausea (Gastrointestinal disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Neuralgia (Nervous system disorders) | 3 (3) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pain (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Paraesthesia (Nervous system disorders) | 1 (2) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Peroneal nerve palsy (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Post procedural infection (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Prostate infection (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Pruritis (Skin and subcutaneous tissue disorders) | 5 (5) — Three subjects adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue. Two subjects AE were judged to be possibly related to treatment with StrataGraft skin tissue.
Pyrexia (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Oedema (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Oedema peripheral (General disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) — Adverse events (AE) were judged to be probably related to treatment with StrataGraft skin tissue.
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Renal failure, acute (Renal and urinary disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Sarcoidosis (Immune system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Sensory disturbance (Nervous system disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Sepsis (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Sinusitis (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Tachycardia (Cardiac disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Thrombophlebitis (Vascular disorders) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Urinary tract infection (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Wound drainage (Surgical and medical procedures) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.
Wound infection, Staphylococcal (Infections and infestations) | 1 (1) — All adverse events (AE) were judged to be unrelated to treatment with StrataGraft skin tissue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No